CLINICAL TRIAL: NCT03551262
Title: Over-the-scope Clip Versus Through-the-scope Clip for Endoscopic Hemostasis of High Risk Bleeding Peptic Ulcers
Acronym: OTSCvsTTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda USL Modena (Other)
Responsible Party: Principal Investigator, Dr. Mauro Manno, Director, Head of Digestive Endoscopy Unit, Principal Investigator, Azienda USL Modena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-2017
Record Dates: First submitted 2017-10-13; First posted 2018-06-11 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2022-07

CONDITIONS: Bleeding Peptic Ulcer
MeSH Terms: conditions — Peptic Ulcer Hemorrhage

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective, randomized, controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OTSC (Experimental): Use of OTSC to treat high-risk peptic ulcers (gastric and duodenal), i.e. Forrest Ia, Ib, IIa, IIb, in first-line endoscopic haemostatic treatment.
  Interventions: Device: OTSC
- TTS clip (Active Comparator): Use of TTS clip to treat high-risk peptic ulcers (gastric and duodenal), i.e. Forrest Ia, Ib, IIa, IIb in first-line endoscopic haemostatic treatment
  Interventions: Device: TTS clip

INTERVENTIONS:
Device: OTSC — Positioning of OTSC in bleeding peptic ulcer
  Arms: OTSC
Device: TTS clip — Positioning of TTS clip in bleeding peptic ulcer
  Arms: TTS clip

SUMMARY:
To compare in a multicenter, prospective, randomized, controlled trial the efficacy and safety of OTSC versus TTS clip for first-line hemostasis of high risk bleeding peptic ulcers

DETAILED DESCRIPTION:
Despite major advances in the management of non-variceal upper gastrointestinal bleeding (NVUGIB) over the past decade including prevention of peptic ulcer bleeding, optimal use of endoscopic therapy and high-dose proton pump inhibition, this still carries considerable morbidity, mortality and health economic burden Of particular note are the re-bleeding rates, one of the most crucial predictive factors of morbidity and mortality that has not significantly improved as evident from longitudinal data in the past 15 years Although huge advances have been made in terms of therapeutic endoscopic devices available today, complete haemostasis of complicated lesions (i.e. severe bleeding from large vessels or fibrotic ulcer) still remains a challenge and can be difficult to achieve. In particular, traditional clipping devices often appear technically difficult to place and insufficient to provide adequate tissue compression to obliterate large bleeding vessels.

The over-the-scope clip (OTSC) (Ovesco Endoscopy AG, Tubingen, Germany) system is a recently developed endoscopic device. In a preliminary experience, it has been successfully used in patients with severe bleeding or deep wall lesions, or perforations of the GI tract.

Recent retrospectives studies have demonstrated the efficacy and safety of OTSC in patients undergoing emergency endoscopy for severe acute NVUGIB after failure of conventional techniques and as first-line To the best of the investigator's knowledge, no randomized clinical trial have been performed investigating the use of OTSC as first-line endoscopic treatment in patients with high-risk NVUGIB.

ELIGIBILITY:
Inclusion Criteria:

* patients with suspected NVUGIB and subsequent endoscopic finding of peptic ulcer (Ia-IIb according to Forrest classification)
* age ≥ 18 years

Exclusion Criteria:

* patients who refused to participate at the trial
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2018-10-26 (Actual); Primary Completion 2023-10-26 (Estimated); Study Completion 2023-10-26 (Estimated)

PRIMARY OUTCOMES:
successful haemostasis rate | during the EGDS
  defined as the absence of bleeding upon at least one minute observation after the assigned endoscopic therapy
30-day rebleeding | up to 30 days
  re-bleeding episodes (per patient), after the primary endoscopic hemostatic treatment, defined as one or more of the following signs:
  * hematemesis
  * presence of fresh blood in the nasogastric tube
  * hemodynamic instability (pulse and blood pressure)
  * reduction of Hb by more than 2 g/dL over a 24 h period (early recurrence) or over a 7 days period (late recurrence) after initial stabilization
overall clinical success | up to 30 days
  defined as successful homeostasis rate without evidence of 30-day rebleeding

SECONDARY OUTCOMES:
mortality | up to 30 days
  number of patients dead with no more rebleeding episodes and number of patients dead with rebleeding episodes, despite the endoscopic treatment
lenght of hospital stay | up to 30 days
  number of days during the hospital stay
transfusion requirements | up to 30 days
  number of transfunsions needed
need for radiology | up to 30 days
  further radiological procedure because of the previous endoscopic failure
need for surgery | up to 30 days
  further surgical procedure because of the previous endoscopic and radiological failures

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Manno, MD, Principal Investigator — Digestive Endoscopy Unit, Northen Area, AUSL Modena (Italy)
Locations (1):
- Azienda USL Modena, Carpi, Modena, Italy

IPD SHARING:
Plan to Share IPD: No